CLINICAL TRIAL: NCT03992235
Title: Importance of Exercise Educational Materials in Chest Physiotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, esra pehlivan, Ass.Prof, PT, PhD, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Educational material
Record Dates: First submitted 2019-06-18; First posted 2019-06-20 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Educational Problems; Physiotherapy; Chest Physiotherapy
Keywords: chest physiotherapy; physiotherapy; education; educational material; thoracotomy; chest; surgery; lung; exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: The patients will randomize into 2 group
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Chest physiotherapy + educational material
  Interventions: Other: Chest physiotherapy; Other: Educational material
- Control group (Other): Chest physiotherapy
  Interventions: Other: Chest physiotherapy

INTERVENTIONS:
Other: Chest physiotherapy — All patients will receive chest physiotherapy including "Breathing exercise, intensive spirometry use, coughing, ambulation".
Other: Educational material — Exercise brochure with photos and explanations
  Arms: Study Group

SUMMARY:
The patients who have undergone thoracotomy operation will include in the study. All patients have chest physiotherapy in the intensive care unit. Patients will be randomized and divided into two groups. One group will be given an exercise form with details and photographs of the exercises. No documents will be given to the other group. The program includes breathing exercises, incentive spirometry study, coughing and graded ambulation. After 1 intensive care session, patients are admitted to the service rooms due to routine procedures. The patients will be served in the afternoon and will be questioned whether they are performing their exercises or not.

DETAILED DESCRIPTION:
* Physiotherapy will be applied to patients undergoing thoracotomy after 24 hours of intensive care hospitalization.
* Patients will be randomized and divided into two groups. Study group will be given exercise form. Control group not.
* Physiotherapy program includes breathing exercises, incentive spirometry study, graded ambulation and both groups will receive this physiotherapy session in the intensive care unit..
* After the patients are admitted to the service rooms, a service visit will be performed, the amount of remembering of the exercises and whether the exercises are performed in a proper form will be questioned.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-70 years
* Having undergone post-thoracotomy
* Hemodynamically stable,
* To be conscious

Exclusion Criteria:

* Excessive pain
* Neurological complications
* Cardiovascular and musculoskeletal problems that prevent him from exercising
* Not wanting to be involved in the study
* Fever above 38 degrees

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
The number of exercises remembered | 15 second
  The number of remembered exercises will be asked by the patient to show the exercises and recorded by the physiotherapist.
The number of exercises done correctly | 15 second
  The number of exercises done correctly will be asked by the patient to show the exercises and recorded by the physiotherapist.

SECONDARY OUTCOMES:
Demographic features | 5 second
  Patients demographic features will be ask to patient

CONTACTS AND LOCATIONS:
Overall Officials: ESRA PEHLİVAN, PhD, Principal Investigator — SBÜ
Locations (1):
- Yedikule Chest Disease Hospital, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No